CLINICAL TRIAL: NCT01757873
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Z160 in Subjects With Postherpetic Neuralgia
Brief Title: Efficacy and Safety Study of Z160 in Subjects With Postherpetic Neuralgia
Acronym: PHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z160-PHN-202
Record Dates: First submitted 2012-12-07; First posted 2012-12-31 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Z160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Z160 (Experimental): 375 mg BID
  Interventions: Drug: Z160
- Placebo (Placebo Comparator): matching placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Z160
  Arms: Z160
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will compare Z160 and placebo in patients with Postherpetic Neuralgia for safety and efficacy for a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Either sex but must be aged >=18 years.
* Diagnosis of PHN as defined by the presence of pain in the area affected by herpes zoster >=6 months after the herpes zoster skin rash has healed.
* Pain score over the last week of >=3 and <=8 on the PI-NRS
* If female, the subject must be postmenopausal , surgically sterilized for >=3 months before the screening visit, or agree to use 2 reliable methods of contraception if of childbearing potential. If male, the subject must agree to use condoms.
* Willing and able to comply with all study procedures.

Exclusion Criteria:

* Severe pain caused by diseases other than PHN.
* Neurolytic or neurosurgical therapy for PHN within 6 months of screening (subjects who received a spinal cord stimulator implant at least 6 months before screening are eligible, but the settings need to remain stable during the double blind study period without use of a magnet).
* History of seizure, excluding pediatric febrile seizures, or currently has seizures.
* Stroke or transient ischemic attack (TIA) <=6 months before the screening visit.
* History of or a current diagnosis of schizophrenia or bipolar disorder.
* Major depressive disorder or generalized anxiety disorder <=6 months before the screening visit. Subjects who are on stable doses of selective serotonin uptake inhibitors (SSRIs) for depression (other than major depressive disorder) are eligible for the study.
* Clinically significant alcohol or substance dependency <=1 year before the screening visit
* Imminent risk of suicide (positive response to question 4 or 5 on the C-SSRS) or had a suicide attempt within 6 months before the screening visit.
* Clinically significant conditions that, in the investigator's opinion, may interfere with the study procedures or compromise the subject's safety.
* Malignancy (other than nonmetastatic basal or squamous cell carcinoma of the skin or carcinoma in situ of other organs that was surgically removed >1 year before screening and has not recurred).
* Condition that is known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Illness within 30 days before screening.
* History of hypersensitivity to calcium channel blockers.
* Multiple drug allergies
* Opioids (at doses exceeding the equivalent of 15 mg of oral morphine) or a high-dose capsaicin patch (Qutenza) <=30 days before the screening visit.
* Moderate or strong cytochrome P450 inducer within 30 days before the screening visit.
* Digoxin or prohibited medications that cannot be discontinued before randomization.
* Other exclusions apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 6 in the weekly average pain score based on Pain Intensity-Numeric Rating Scale (PI-NRS) | Baseline to Week 6

SECONDARY OUTCOMES:
Change from baseline in weekly average pain score | Baseline to Weeks 1, 2, 3, 4, 5, 6
Neuropathic Pain Scale (NPS) | Baseline to Weeks 1, 2, 4, 6
Patient Global Impression of Change (PGIC) | Baseline to Week 6
Profile of Mood States (POMS) | Baseline to Weeks 1, 2, 4, 6
Daily Sleep Interference Scale (DSIS) | Baseline to Weeks 1, 2, 3, 4, 5, 6
Short Form 36 (SF-36) | Baseline to Week 6
Z160 plasma concentrations | Baseline to Weeks 1, 2, 4, 6
Time to a >= 30% reduction in weekly average pain score | Baseline to Weeks 1, 2, 3, 4, 5, 6
Time to a >= 50% reduction in weekly average pain score | Baseline to Weeks 1, 2, 3, 4, 5, 6
Subjects who have >= 30% reduction in average daily pain score | Baseline to Week 6
Subjects who have >= 50% reduction in average daily pain score | Baseline to Week 6
Safety and tolerability | Baseline to Weeks 1- 12
  As measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events
Amount of rescue medication used | Baseline to Weeks 1, 2, 4 and 6

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, Chandler, Arizona
  - Investigative Site, Mesa, Arizona
  - Investigative Site, Peoria, Arizona
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Scottsdale, Arizona
  - Investigative Site, Little Rock, Arkansas
  - Investigative Site, Irvine, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, San Francisco, California
  - Investigative Site, Thousand Oaks, California
  - Investigative Site, Boulder, Colorado
  - Investigative Site, Colorado Springs, Colorado
  - Investigative Site, Denver, Colorado
  - Investigative Site, Brooksville, Florida
  - Investigative Site, Clearwater, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Port Orange, Florida
  - Investigative Site, Royal Palm Beach, Florida
  - Investigative Site, Sarasota, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Evansville, Indiana
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Columbia, Maryland
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Ann Arbor, Michigan
  - Investigative Site, Bay City, Michigan
  - Investigative Site, Ocean Springs, Mississippi
  - Investigative Site, Hazelwood, Missouri
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Toms River, New Jersey
  - Investigative Site, Albuquerque, New Mexico
  - Investigative Site, Brooklyn, New York
  - Investigative Site, New York, New York
  - Investigative Site, Greensboro, North Carolina
  - Investigative Site, Beavercreek, Ohio
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Kettering, Ohio
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Charleston, South Carolina
  - Investigative Site, Nashville, Tennessee
  - Investigative Site, Tullahoma, Tennessee
  - Investigative Site, Austin, Texas
  - Investigative Site, Richardson, Texas
  - Investigative Site, Murray, Utah
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, Herndon, Virginia
  - Investigative Site, Bellevue, Washington
  - Investigative Site, Tacoma, Washington